CLINICAL TRIAL: NCT04478968
Title: The Levels of Fibrosis Biomarkers in Patients After Renal Transplantation in Relation to Arteriovenous Fistula Function
Brief Title: Approach to Vascular Access After Renal Transplantation
Acronym: AVART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MINI.C160.20.001
Record Dates: First submitted 2020-06-29; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-06

CONDITIONS: Kidney Transplantation
Keywords: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active AVF: Patients after kidney transplantation with functioning AVF
  Interventions: Other: presence of AVF
- No AVF: Patients after kidney transplantation without AVF (thrombosed AVF, history of HD with catheter, history of PD, preemptive transplantation)

INTERVENTIONS:
Other: presence of AVF — Functioning AVF may have cardiotoxic potential
  Groups: Active AVF

SUMMARY:
The aim of the project is to assess the effect of functioning AVF in renal transplant patients on fibrosis, inflammation and LVH indicators. Clinical and laboratory parameters will be compared in a group of 150 patients, 75 patients with a functioning fistula and 75 patients with inactive vascular access. We will assess the impact of functional AVF and the levels of biomarkers on the survival of patients and transplanted kidneys.

DETAILED DESCRIPTION:
Patients after kidney transplantation during a routine visit will be asked to participate to the study. In eligible a number of studies will be conducted:

* detailed clinical examination
* routine laboratory tests
* lung ultrasound
* muscle strength with a dynamometer
* ultrasound assessment of upper limb vessels with assessment of fistula function (in the case of active fistula) and for the possibility of future vascular access
* blood collection and protection (10-15 ml) for biomarkers
* survey EQ-5D-5L and LVD-36
* functional strength test.

The obtained clinical data and test results will be subject to statistical analysis after anonymization. The impact of individual parameters on long-term prognosis will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years old
* kidney transplant
* >12 months after transplantation
* stable transplanted kidney function
* signed informed consent

Exclusion Criteria:

* GFR <15 ml / min
* severe infection within 3 months of testing
* increase in creatinine concentration> 0.5 mg / dl within 3 months before the test
* active cancer
* signs of severe heart failure (NYHA IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a kidney transplant belong to the group of patients at increased risk for cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-01-02 (Estimated); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life with EQ-5D-5L | Baseline visit up to 12 months
  The survey results will be compared between the study and control groups to see if the presence of the arteriovenous fistula affects quality of life.
Prognostic value of biomarkers (NT-proBNP, Il-6, sST2, galectin-3, GDF-15, MMP7, TIMP1) | Baseline visit and up to 12 months
  The levels of biomarkers will be measured and the results will be compared between the study and control groups. A prognostic value of the biomarkers will be estimated.

SECONDARY OUTCOMES:
Hospitalization-free survival | Up to 12 months from baseline visit
  Hospital-free survival will be reported as the number of patients living 12 months after the initial visit without the need for hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Letachowicz, MD, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Department of Nephrology and Transplantation Medicine, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided